CLINICAL TRIAL: NCT05767788
Title: Effectiveness of Mobilization With Movement (MWM) on Patients With Knee Osteoarthritis (OA): A Double-blinded Randomized Sham-controlled Trial
Brief Title: Mobilization With Movement (MWM) on Knee Osteoarthritis (OA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MWMKOA
Record Dates: First submitted 2023-01-31; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Movement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Movement with Mobilization (MWM) (Experimental): Active movement with passive mobilization gliding force
  Interventions: Other: Movement with Mobilization (MWM)
- Sham Movement with Mobilization (Sham MWM) (Sham Comparator): Active movement with passive light touch gliding force
  Interventions: Other: Sham Movement with Mobilization (Sham MWM)

INTERVENTIONS:
Other: Movement with Mobilization (MWM) — Painful active functional knee movement is identified. The most comfortable passive medial, lateral, medial rotatory, lateral rotatory, postero-anterior, and antero-posterior glide, is applied to the knee of the patient.
  Three sets of 10 repetitions are applied. Corresponding home MWM exercise is taught. The treatment is conducted for 12 sessions over 6 weeks.
  Arms: Movement with Mobilization (MWM)
Other: Sham Movement with Mobilization (Sham MWM) — Painful active functional knee movement is identified. The most comfortable passive medial, lateral, medial rotatory, lateral rotatory, postero-anterior, and antero-posterior light-touch glide, is applied to the knee of the patient.
  Three sets of 10 repetitions are applied. Corresponding home MWM exercise is taught. The treatment is conducted for 12 sessions over 6 weeks.
  Arms: Sham Movement with Mobilization (Sham MWM)

SUMMARY:
Movement with mobilization (MWM) is an effective manual therapy to improve pain and function of patients with knee osteoarthritis (OA).

However, immediate, and prolonged effects after prolonged MWM period was under-investigated.

In this double-blinded randomized control trial, 40 patients are needed. The subjects and assessors will be blinded. Subjects in intervention group will receive MWM twice a week and corresponding home exercise for 6 weeks.

Participants in control group will only receive sham treatment with light touch.

The effects on knee pain in visual analogue scale (VAS); flexion and extension range of motion (ROM) by goniometer; strength by hand-held dynamometer; function by Timed Up and Go Test (TUG) and 30-second Chair Stand Test; and health-related quality of life (HRQoL) by Knee Injury and Osteoarthritis Outcome Score (KOOS) and Western Ontario and McMaster Universities Arthritis Index (WOMAC) just after, 1-month and 3-month after treatment will be compared with baseline. Six-month after treatment, KOOS and WOMAC will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* History of knee OA for at least 1-year
* Pain intensity level ≥ 3 on a 10-cm Visual Analogue Scale (VAS)
* Both unilateral or bilateral knee pain
* Having morning stiffness less than 30 minutes
* Having crepitus on active movement
* Having bony tenderness
* Having bony enlargement

Exclusion Criteria:

* Having active inflammatory or infectious knee conditions
* Having bone integrity conditions like osteoporosis
* Having knee joint instability
* Having skin integrity conditions like frail skin or lower limb peripheral vascular disease
* History of hip or knee fracture
* History of knee surgical history
* Use of knee corticosteroid or opioid injection

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-05-10 (Estimated); Study Completion 2023-05-10 (Estimated)

PRIMARY OUTCOMES:
Change of pain in the Visual Analogue Scale (VAS) | The change before the start of treatment and after 6-week treatment
  Subjects will indicate the pain level on a 100-millimeter line with endpoints, marked "no pain" and "worst imaginable pain", at the time of assessment.
Change of pain in the Visual Analogue Scale (VAS) | The change before the start of treatment and 1-month after last treatment session
  Subjects will indicate the pain level on a 100-millimeter line with endpoints, marked "no pain" and "worst imaginable pain", at the time of assessment.
Change of pain in the Visual Analogue Scale (VAS) | The change before the start of treatment and 3-month after last treatment session
  Subjects will indicate the pain level on a 100-millimeter line with endpoints, marked "no pain" and "worst imaginable pain", at the time of assessment.

SECONDARY OUTCOMES:
Change of time used in the Timed Up and Go Test (TUG) | The change before the start of treatment and after 6-week treatment
  Subjects will be instructed to get up from the chair and then walk to a target 3 meters away, turn around, walk back to the chair, and sit down. The time used will be recorded. An average of two testing trials will be used.
Change of time used in the Timed Up and Go Test (TUG) | The change before the start of treatment and 1-month after last treatment session
  Subjects will be instructed to get up from the chair and then walk to a target 3 meters away, turn around, walk back to the chair, and sit down. The time used will be recorded. An average of two testing trials will be used.
Change of time used in the Timed Up and Go Test (TUG) | The change before the start of treatment and 3-month after last treatment session
  Subjects will be instructed to get up from the chair and then walk to a target 3 meters away, turn around, walk back to the chair, and sit down. The time used will be recorded. An average of two testing trials will be used.
Change of number of repetitions in the 30-second Chair Stand Test (30CST) | The change before the start of treatment and after 6-week treatment
  Subjects will be instructed to stand up from the chair and then return to sit down on the chair repeatedly for 30 seconds or until the subject fails to continue at any time point during the trial. Only 1 testing trial will be used.
Change of number of repetitions in the 30-second Chair Stand Test (30CST) | The change before the start of treatment and 1-month after last treatment session
  Subjects will be instructed to stand up from the chair and then return to sit down on the chair repeatedly for 30 seconds or until the subject fails to continue at any time point during the trial. Only 1 testing trial will be used.
Change of number of repetitions in the 30-second Chair Stand Test (30CST) | The change before the start of treatment and 3-month after last treatment session
  Subjects will be instructed to stand up from the chair and then return to sit down on the chair repeatedly for 30 seconds or until the subject fails to continue at any time point during the trial. Only 1 testing trial will be used.
Change of knee flexors muscle strength by the hand-held dynamometer | The change before the start of treatment and after 6-week treatment
  A digital dynamometer will be used to measure the muscle strength (in kilograms) of the subject's hamstrings muscles. Subjects will be guided to sit with their arms crossed at the shoulders and hold against their chest, back straight, knees relax in 90 degrees flexion in a high sitting position. The isometric peak force for flexion will be recorded respectively.
  An average of 3 testing trials will be used.
Change of knee flexors muscle strength by the hand-held dynamometer | The change before the start of treatment and 1-month after last treatment session
  A digital dynamometer will be used to measure the muscle strength (in kilograms) of the subject's hamstrings muscles. Subjects will be guided to sit with their arms crossed at the shoulders and hold against their chest, back straight, knees relax in 90 degrees flexion in a high sitting position. The isometric peak force for flexion will be recorded respectively.
  An average of 3 testing trials will be used.
Change of knee flexors muscle strength by the hand-held dynamometer | The change before the start of treatment and 3-month after last treatment session
  A digital dynamometer will be used to measure the muscle strength (in kilograms) of the subject's hamstrings muscles. Subjects will be guided to sit with their arms crossed at the shoulders and hold against their chest, back straight, knees relax in 90 degrees flexion in a high sitting position. The isometric peak force for flexion will be recorded respectively.
  An average of 3 testing trials will be used.
Change of knee extensors muscle strength by the hand-held dynamometer | The change before the start of treatment and after 6-week treatment
  A digital dynamometer will be used to measure the muscle strength (in kilograms) of the subject's quadriceps and muscles.
  Subjects will be guided to sit with their arms crossed at the shoulders and hold against their chest, back straight, knees relax in 90 degrees flexion in a high sitting position.
  The isometric peak force for flexion and extension will be recorded respectively.
  An average of 3 testing trials will be used.
Change of knee extensors muscle strength by the hand-held dynamometer | The change before the start of treatment and 1-month after last treatment session
  A digital dynamometer will be used to measure the muscle strength (in kilograms) of the subject's quadriceps and muscles.
  Subjects will be guided to sit with their arms crossed at the shoulders and hold against their chest, back straight, knees relax in 90 degrees flexion in a high sitting position.
  The isometric peak force for flexion and extension will be recorded respectively.
  An average of 3 testing trials will be used.
Change of knee extensors muscle strength by the hand-held dynamometer | The change before the start of treatment and 3-month after last treatment session
  A digital dynamometer will be used to measure the muscle strength (in kilograms) of the subject's quadriceps and muscles.
  Subjects will be guided to sit with their arms crossed at the shoulders and hold against their chest, back straight, knees relax in 90 degrees flexion in a high sitting position.
  The isometric peak force for flexion and extension will be recorded respectively.
  An average of 3 testing trials will be used.
Change of score of the Knee Injury and Osteoarthritis Outcome Score (KOOS) | The change before the start of treatment and after 6-week treatment
  A health-related quality of life questionnaire. The score ranges from 0% (the worst) to 100% (the best).
Change of score of the Knee Injury and Osteoarthritis Outcome Score (KOOS) | The change before the start of treatment and 1-month after last treatment session
  A health-related quality of life questionnaire. The score ranges from 0% (the worst) to 100% (the best).
Change of score of the Knee Injury and Osteoarthritis Outcome Score (KOOS) | The change before the start of treatment and 3-month after last treatment session
  A health-related quality of life questionnaire. The score ranges from 0% (the worst) to 100% (the best).
Change of score of the Knee Injury and Osteoarthritis Outcome Score (KOOS) | The change before the start of treatment and 6-month after last treatment session
  A health-related quality of life questionnaire. The score ranges from 0% (the worst) to 100% (the best).
Change of score of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) | The change before the start of treatment and after 6-week treatment
  A health-related quality of life questionnaire. The score ranges from 0 (the worst) to 100 (the best).
Change of score of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) | The change before the start of treatment and 1-month after last treatment session
  A health-related quality of life questionnaire. The score ranges from 0 (the worst) to 100 (the best).
Change of score of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) | The change before the start of treatment and 3-month after last treatment session
  A health-related quality of life questionnaire. The score ranges from 0 (the worst) to 100 (the best).
Change of score of the Western Ontario and McMaster Universities Arthritis Index (WOMAC) | The change before the start of treatment and 6-month after last treatment session
  A health-related quality of life questionnaire. The score ranges from 0 (the worst) to 100 (the best).
Change of active knee flexion range of motion by the standard goniometer | The change before the start of treatment and after 6-week treatment
  The active range of motion for knee flexion will be measured with a standard goniometer on the painful knee in supine.
  An average of 3 testing trials will be used.
Change of active knee flexion range of motion by the standard goniometer | The change before the start of treatment and 1-month after last treatment session
  The active range of motion for knee flexion will be measured with a standard goniometer on the painful knee in supine.
  An average of 3 testing trials will be used.
Change of active knee flexion range of motion by the standard goniometer | The change before the start of treatment and 3-month after last treatment session
  The active range of motion for knee flexion will be measured with a standard goniometer on the painful knee in supine.
  An average of 3 testing trials will be used.
Change of active knee extension range of motion by the standard goniometer | The change before the start of treatment and after 6-week treatment
  The active range of motion for knee flexion will be measured with a standard goniometer on the painful knee in supine.
  An average of 3 testing trials will be used.
Change of active knee extension range of motion by the standard goniometer | The change before the start of treatment and 1-month after last treatment session
  The active range of motion for knee flexion will be measured with a standard goniometer on the painful knee in supine.
  An average of 3 testing trials will be used.
Change of active knee extension range of motion by the standard goniometer | The change before the start of treatment and 3-month after last treatment session
  The active range of motion for knee flexion will be measured with a standard goniometer on the painful knee in supine.
  An average of 3 testing trials will be used.

CONTACTS AND LOCATIONS:
Overall Officials: KING HIM CHAN, BSc, Principal Investigator — Department of Rehabilitation Sciences, The Hong Kong Polytechnic University; MING HON LEE, BSc, Principal Investigator — Department of Rehabilitation Sciences, The Hong Kong Polytechnic University; YIK SING SHUM, BSc, Principal Investigator — Department of Rehabilitation Sciences, The Hong Kong Polytechnic University; YEUK LAI CHAN, BSc, Principal Investigator — Department of Rehabilitation Sciences, The Hong Kong Polytechnic University; FADI AL ZOUBI, PhD, Principal Investigator — Department of Rehabilitation Sciences, The Hong Kong Polytechnic University; MAN HA TSANG, PhD, Principal Investigator — Department of Rehabilitation Sciences, The Hong Kong Polytechnic University
Locations (1):
- Department of Rehabilitation Sciences, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided